CLINICAL TRIAL: NCT02679001
Title: A COMPARATIVE OBSERVATIONAL STUDY FOLLOWING THE USE OF CONCOMITANT CORTICOSTEROID TREATMENT IN RA PATIENTS WHO ARE TREATED WITH A TNF INHIBITOR OR TOCILIZUMAB AS THEIR SECOND BIOLOGICAL TREATMENT
Brief Title: A Comparative Study to Observe the Effect of Concomitant Use of Corticosteroid Treatment in Rheumatoid Arthritis (RA) Participants Who Are Treated With a Tumor Necrosis Factor (TNF) Inhibitor or Tocilizumab (TCZ) as Their Second Biological Treatment.
Status: Completed | Type: Observational
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Other Study IDs: ML29933
Record Dates: First submitted 2016-02-08; First posted 2016-02-10 (Estimated); Last update posted 2018-07-26 (Actual); Status verified 2018-07

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional

GROUPS / COHORTS (1):
- RA participants treated with a TNF inhibitor or TCZ: Participants with RA receiving TNF-inhibitor or TCZ according to standard of care and in line with the current summary of product characteristics (SPC)/local labeling will be observed.
  Interventions: Drug: TNF inhibitor/TCZ

INTERVENTIONS:
Drug: TNF inhibitor/TCZ — Participants with RA receiving TNF-inhibitor or TCZ according to standard of care and in line with the current SPC/local labeling will be observed.
  Other Names: COTTON

SUMMARY:
This six months non-interventional, observational, post-marketing, multi-center and local study will evaluate the differences in the use of corticosteroids between RA participants receiving TCZ or a TNF-inhibitor, in participants who have discontinued the use of a TNF-inhibitor as their first biological treatment.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age.
* With a diagnosis of moderate to severe RA according to the revised (1987) American College of Rheumatology (ACR) criteria or 2010 ACR/ European League Against Rheumatism (EULAR) RA classification criteria.
* Have had an insufficient response or intolerance to their first TNF-inhibitor (including biosimilars for TNF-inhibitors).
* The treating physician has made the decision to commence TCZ or TNF-inhibitor treatment. Participants need to have a Disease Activity Score (DAS) 28 assessment at initiation of their second biological treatment.
* Have been given oral and written information about the study and have no objection to the data concerning him/her being subject to computerized data processing, have given informed consent.

Exclusion Criteria:

* Have had more than one TNF-inhibitor prior to the enrolment visit.
* Have had biological treatment other than TNF-inhibitors.
* Participants that are continuously treated with per oral corticosteroids for any other indication than RA (at baseline).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants with a diagnosis of moderate to severe RA according to the revised (1987) ACR criteria or 2010 ACR/EULAR RA classification criteria who have had an insufficient response or intolerance to their first TNF-inhibitor.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2016-03-24 (Actual); Primary Completion 2017-12-07 (Actual); Study Completion 2017-12-07 (Actual)

PRIMARY OUTCOMES:
Percentage of participants with a decrease in dose of oral corticosteroids during the study | From baseline to 6 months

SECONDARY OUTCOMES:
Percentage of participants achieving C59CDAI remission (</=2.8) | From baseline to 6 months
Percentage of participants achieving CDAI LDA (</=10) | From baseline to 6 months
Percentage of participants using non-biologic disease-modifying anti-rheumatic drugs (C58MARDs) at treatment initiation and at the end of observation period | Baseline, Month 6
Percentage of participants for whom non-biologic DMARDs was added during observation period | From baseline to 6 months
Percentage of participants with dose change in biological treatment during study | From baseline to 6 months
Percentage of participants with use of oral corticosteroids at treatment initiation and at end of study | From baseline to 6 months
Percentage of participants who started or stopped oral corticosteroid treatment during the study period | From baseline to 6 months
Percentage of participants with increased/decreased/stable dose of corticosteroids from baseline to end of study | From baseline to 6 months
Percentage of participants with change in dose of corticosteroids during study but with same dose at study end as at baseline | From baseline to 6 months
Cumulated doses of oral corticosteroids during study period | From baseline to 6 months
Number of corticosteroids including but not limited to intra-articular, intravenously, inhaled, topical and/or intramuscular/subcutaneous injections | From baseline to 6 months
Cumulated doses of corticosteroids including but not limited to intra-articular, intravenously, inhaled, topical and/or intramuscular/subcutaneous injections | From baseline to 6 months
Cumulated doses of all corticosteroids during study period | From baseline to 6 months
Mean dose of corticosteroids at start and end of study | From baseline to 6 months
Mean change from baseline to end of study of corticosteroids | Baseline, Month 6
Mean change from baseline to end of study in DAS28 (sedimentation rate [SR]) score | Baseline, Month 6
Mean change from baseline to end of study in DAS28 (C-Reactive Protein [CRP]) score | Baseline, Month 6
Mean change from baseline to end of study in crohns disease activity index (CDAI) score | Baseline, Month 6
Mean change from baseline to end of study in swollen 28 joint count | Baseline, Month 6
Mean change from baseline to end of study in tender 28 joint count | Baseline, Month 6
Mean change from baseline to end of study in Physician Global Assessment of disease activity (Visual Analogue Scale [VAS] scale) | Baseline, Month 6
Mean change from baseline to end of study in Patient Global Assessment of disease activity (VAS scale) | Baseline, Month 6
Mean change from baseline to end of study in Health Assessment Questionnaire Disability Index (HAQ-DI) | Baseline, Month 6
Mean change from baseline to end of study in Severity of pain (VAS scale) | Baseline, Month 6
Mean change from baseline to end of study in EULAR response | Baseline, Month 6
Percentage of participants achieving DAS28 remission (less than or equal to [</=] 2.6) | From baseline to 6 months
Percentage of participants achieving DAS 28 Low Disease Activity (LDA) (</=3.2) | From baseline to 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (11):
- Sweden (11):
  - Arvika Sjukhus; Reumatologimottagningen - Medicinmottagningen, Arvika
  - Mälarsjukhuset; Reumatologkliniken, Eskilstuna
  - Karolinska University Hospital, Huddinge; Rheumatology, Huddinge
  - Blekingesjukhuset Karlskrona; Medicin, Rheumatology, Karlskrona
  - Skånes Universitetssjukhus Malmö; Reumatologkliniken, Malmo
  - Capio Citykliniken, Reumatologen, Malmo
  - Örebro Uni Hospital; Rheumatology, Örebro
  - Kaernsjukhuset; Dept of Medicine, Skövde
  - Danderyds Sjukhus Ab; Rheumatology, Stockholm
  - Lasarettet Trelleborg;Reumatologmottagningen, Trelleborg
  - Akademiska sjukhuset, Reumatologkliniken, Uppsala